CLINICAL TRIAL: NCT05708898
Title: Effect of Pharyngeal Exerciser in Rehabilitation of Pharyngeal Phase of Swallowing in Patients With Dysphagia
Brief Title: External Pharyngeal Exerciser and Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Reza Shaker, MD, Associate Provost for Clinical and Translational Research, Senior Associate Dean and Director of the Clinical and Translational Science Institute of SE WI, and the Joseph E. Geenen Professor and Chief of Gastroenterology and Hepatology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00023967
Record Dates: First submitted 2023-01-13; First posted 2023-02-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Pharyngeal exerciser group: In this group, the device will be placed around the neck overlying the laryngeal cartilage using the Velcro fastening in the back of neck. The externally applied pressure will be measured via the pressure gauge included in the device (see figure). Patients are asked to follow exercise regimen: to perform 30 swallows at 15 seconds interval against minimal resistance of 20 mm Hg applied by pharyngeal exerciser over larynx during the first 2 weeks. This is repeated 3 times per day and the external resistance is increased every 2 weeks from 20 to 30 mm Hg and subsequently from 30 to 40 mm Hg in another 2 weeks.
  Sham exerciser group: In this group, sham device will be placed around the neck overlying the laryngeal cartilage. No external pressure will be applied during exercise. These patients will be asked to follow the exercise regimen: to perform repetitive tongue protrusion for 5 times without any pressure. This will be repeated 3 times a day for 6 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Pharyngeal exerciser group (Experimental): In this group, the device will be placed around the neck overlying the laryngeal cartilage. Patients are asked to follow exercise regimen: to perform 30 swallows at 15 seconds interval against minimal resistance of 20 mm Hg applied by pharyngeal exerciser over larynx during the first 2 weeks. This is repeated 3 times per day and the external resistance is increased every 2 weeks from 20 to 30 mm Hg and subsequently from 30 to 40 mm Hg in another 2 weeks.
  Interventions: Device: Pharyngeal exerciser
- Sham exerciser group (Sham Comparator): In this group, sham device will be placed around the neck overlying the laryngeal cartilage. No external pressure will be applied during exercise. These patients will be asked to follow the exercise regimen: to perform repetitive tongue protrusion for 5 times without any pressure. This will be repeated 3 times a day for 6 weeks.
  Interventions: Device: sham pharyngeal exerciser

INTERVENTIONS:
Device: Pharyngeal exerciser
  Arms: Pharyngeal exerciser group
Device: sham pharyngeal exerciser
  Arms: Sham exerciser group

SUMMARY:
The goal of this a clinical trial is to test the effect of a pharyngeal exerciser in rehabilitation of pharyngeal phase of swallowing in patients with dysphagia. The main question it aims to answer is:

•Does application of pharyngeal exerciser improve swallowing as evidenced by need for prescribed intervention for dysphagia (maneuvers, exercises or dietary modification to prevent aspiration).

Participants will:

* Perform barium swallows in lateral view fluoroscopy
* Over a six-week period, perform thrice daily sessions of swallowing with an external, laryngeal restriction device covering the larynx
* Return for another fluoroscopic barium swallow study

DETAILED DESCRIPTION:
All the patients will be reviewed for inclusion and exclusion of the study in detailed manner using medical evaluation form. The physical examination part of the medical evaluation form will be filled out by one of our designated physician investigators. A urine pregnancy test will be administered if necessary at this time.

The patient's neck physical dimensions and device's physical dimensions will be measured and recorded using the Biometric form.

A baseline functional outcome assessment of swallowing (FOAMS) will be performed for each patient.

Patients will be sitting in an upright position with the head held in neutral position at Fluoroscopy lab and acclimatized for 10 minutes before proceeding.

Patient's anatomic structure and landmarks are identified in both lateral and anteroposterior (AP) views with fluoroscopy.

A 4 mm diameter catheter with 3 markers 3 cm apart will be placed on the skin in the pharyngo-UES region for the purpose of calibration and nullify the error from magnification during videorecording.

Patient will be asked to swallow barium suspension at incremental volumes of 1, 3 and 5 ml; however, if the patient develops aspiration or doesn't tolerate barium suspension higher volumes will not be administered. Following are test swallows under fluoroscopy:

1 ml- 40% weight/volume barium suspension at room temperature x 3 times each. 3 ml- 40% weight/volume barium suspension at room temperature x 3 times each. 5 ml- 40% weight/volume barium suspension at room temperature x 3 times each. The fluoroscopy machine will be turned "on" for 5 seconds ONLY during each swallow. Rest of the time fluoroscopy machine will be turned "off".

Fluoroscopic recordings were obtained at 90 kilo-electron-volt (KeV), using a 9-inch image-intensifier mode and appropriate collimation so that an image was obtained of the posterior mouth, pharynx, and pharyngoesophageal region. Fluoroscopic recordings will be timed using a specially designed timer.

After the baseline fluoroscopic study, each patient will be randomized to receive either the sham exerciser (i.e. device with no pressure) or pharyngeal exerciser (i.e. device with graded pressure).

Study Groups:

Pharyngeal exerciser group: In this group, the device will be placed around the neck overlying the laryngeal cartilage. The device will be in contact with the skin without any underlying pressure using the Velcro fastening in the back of neck. The externally applied pressure will be measured by means of the pressure gauge included in the device (see figure). Patients are asked to follow exercise regimen: to perform 30 swallows at 15 seconds interval against minimal resistance of 20 mm Hg applied by pharyngeal exerciser over larynx during the first 2 weeks. This is repeated 3 times per day and the external resistance is increased every 2 weeks from 20 to 30 mm Hg and subsequently from 30 to 40 mm Hg in another 2 weeks.

Sham exerciser group: In this group, sham device will be placed around the neck overlying the laryngeal cartilage. No external pressure will be applied during exercise. These patients will be asked to follow the exercise regimen: to perform repetitive tongue protrusion for 5 times without any pressure. This will be repeated 3 times a day for 6 weeks.

All the exercise instructions and log record will be given to each of the patient in both study groups at the time of randomization. The exerciser (sham or pharyngeal) will be worn only at the time of exercises.

Weekly telephone interviews will be conducted to assess their progress and address their concerns in both study groups.

Patients in both study groups are required to make follow up visits every 2 weeks. During the follow up visits, patients will be reviewed for symptom severity and resistance of the device. This information is documented in patient progress sheet and follow up visit form. All the adverse events during the study or from the device will be documented in the adverse and serious adverse events form. The compliance with the device will be evaluated by examining the exercise log sheet.

After 6 weeks, the device (sham exerciser or pharyngeal exerciser) will be returned to the study team and patients will be asked to complete functional outcome assessment of swallowing (FOAMS).

Each patient will undergo follow up fluoroscopic study with the same test swallows as the baseline swallows, looking for pharyngeal residue and aspiration (repeat steps: 4 to 9).

All the fluoroscopic images will be recorded and stored in digitalized format at 30 frames (60 fields/second) in a secure location at the research lab (locked in safe location and accessible only to the investigators). These the fluoroscopic studies will be analyzed for the study parameters as mentioned below by two individuals in a blinded fashion.

At the end of study period, each of the patients in sham group will be given an option to undergo another 6 weeks of pharyngeal exercise using pharyngeal exerciser. If they consent again(using informed consent form) to participate, they would be following above exercise protocol(30 swallows against 20 mm Hg of resistance with pharyngeal exerciser three times a day for 2 weeks; followed by swallowing exercise with incremental resistance of 30 and 40 mm Hg for 2 weeks each). At of 6 weeks, they would undergo repeat fluoroscopy study to check for improvement in pharyngeal residue (repeat steps: 4 to 9).

The participants will be followed after completion of the exercise regimen for a total of 12 months. At 3 months after the completion of initial exercise study, the participant will be contacted and informed about the follow up portion of the study. If they are in agreement, the participant will be asked to come to the lab to be reconsented and complete an EAT-10 form. At this time, the participant will be asked questions such as current diet consistency, evidence of cough with eating, additional time needed during meals, etc to determine FOAMS score. The patient will only be interviewed after consent is obtained. At 6 months, the subjects will undergo repeat fluoroscopy for an objective measure of their swallowing. At this visit they will also be asked to complete an EAT-10 form and a FOAMS score will again be determined. At 12 months, the participant will not be required to return to the lab. They will also be mailed a swallowing assessment form (EAT-10) to be filled out and returned at 12 months (subjects will be asked to complete the paper form for consistency). The participant will also be contacted for a telephone interview to be asked questions such as current diet consistency, evidence of cough with eating, additional time needed during meals, etc to determine FOAMS score. For those subjects who are newly enrolled, re-consent will not occur since there is only one consent form which includes the follow-up information. Newly enrolled subjects will be presented with the follow-up information at the time of initial consent.

During the entire study period, the participant will be instructed to continue their standard of medical care (medications, diet, physical therapy and activity) as suggested by their personnel physician.

All the fluoroscopic studies will be analyzed by two individuals in a blinded fashion.

After the completion of the study, individuals in the sham exerciser group will be given the option of doing exercises using pharyngeal exerciser. If they are interested, consent will be obtained using new consent form before re-enrolling into the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysphagia characterized by persistent pharyngeal residue on fluoroscopic study undergoing rehabilitative intervention (e.g.: exercises, maneuvers or dietary modification) for improving swallowing and preventing aspiration

Healthy elderly adult (≥65 years of age).

Exclusion Criteria:

* Patients younger than 18 years of age.

Patients with recent head and neck cancer (<1 month post-surgery or <3 months post-chemo radiation.

Patients suffering from muscle diseases like muscular dystrophies, myopathies.

Patients with neuro-muscular junction disorders myasthenia gravis, Eaton-Lambert disorders

Patients having history of allergy to lidocaine or barium.

Patients who are pregnant or lactating.

Patients who are medically unstable.

Patients who are unable to apply the exerciser independently or with the help of a caregiver.

Patients who lack cognition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-06-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum anterior hyoid excursion | Before six weeks exerciser regimen
  deglutitive maximum anterior hyoid excursion from resting position measured from fluoroscopic images
maximum anterior hyoid excursion | after six weeks exerciser regimen
  deglutitive maximum anterior hyoid excursion from resting position measured from fluoroscopic images
maximum superior hyoid excursion | Before six weeks exerciser regimen
  deglutitive maximum superior hyoid excursion from resting position measured from fluoroscopic images
maximum superior hyoid excursion | after six weeks exerciser regimen
  deglutitive maximum superior hyoid excursion from resting position measured from fluoroscopic images
maximum anterior laryngeal excursion | Before six weeks exerciser regimen
  deglutitive maximum anterior laryngeal excursion from resting position measured from fluoroscopic images
maximum anterior laryngeal excursion | after six weeks exerciser regimen
  deglutitive maximum anterior laryngeal excursion from resting position measured from fluoroscopic images
maximum superior laryngeal excursion | before six weeks exerciser regimen
  deglutitive maximum superior laryngeal excursion from resting position measured from fluoroscopic images
maximum superior laryngeal excursion | after six weeks exerciser regimen
  deglutitive maximum superior laryngeal excursion from resting position measured from fluoroscopic images
maximum upper esophageal sphincter (UES) anterior-posterior opening | Before six weeks exerciser regimen
  deglutitive maximum UES diameter measured from fluoroscopic images
maximum upper esophageal sphincter (UES) anterior-posterior opening | after six weeks exerciser regimen
  deglutitive maximum UES diameter measured from fluoroscopic images
pyriform sinus residue | Before six weeks exerciser regimen
  area (height x width) of pyriform sinus residue measure from fluoroscopic images
pyriform sinus residue | after six weeks exerciser regimen
  area (height x width) of pyriform sinus residue measure from fluoroscopic images

SECONDARY OUTCOMES:
Penetration and aspiration analyses | Before six weeks exerciser regimen
  Reduction of aspiration and penetration measured by Rosenbek's penetration-aspiration scale
Penetration and aspiration analyses | after six weeks exerciser regimen
  Reduction of aspiration and penetration measured by Rosenbek's penetration-aspiration scale

CONTACTS AND LOCATIONS:
Overall Officials: Reza Shaker, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabre M, Serra-Prat M, Palomera E, Almirall J, Pallares R, Clave P. Prevalence and prognostic implications of dysphagia in elderly patients with pneumonia. Age Ageing. 2010 Jan;39(1):39-45. doi: 10.1093/ageing/afp100. Epub 2009 Jun 26. PMID 19561160
- [Background] Turley R, Cohen S. Impact of voice and swallowing problems in the elderly. Otolaryngol Head Neck Surg. 2009 Jan;140(1):33-6. doi: 10.1016/j.otohns.2008.10.010. PMID 19130958
- [Background] Bonilha HS, Simpson AN, Ellis C, Mauldin P, Martin-Harris B, Simpson K. The one-year attributable cost of post-stroke dysphagia. Dysphagia. 2014 Oct;29(5):545-52. doi: 10.1007/s00455-014-9543-8. Epub 2014 Jun 20. PMID 24948438
- [Background] Altman KW, Yu GP, Schaefer SD. Consequence of dysphagia in the hospitalized patient: impact on prognosis and hospital resources. Arch Otolaryngol Head Neck Surg. 2010 Aug;136(8):784-9. doi: 10.1001/archoto.2010.129. PMID 20713754
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Altman KW, Schaefer SD, Yu GP, Hertegard S, Lundy DS, Blumin JH, Maronian NC, Heman-Ackah YD, Abitbol J, Casiano RR; Neurolaryngology Subcommittee of the American Academy of Otolaryngology-Head and Neck Surgery. The voice and laryngeal dysfunction in stroke: a report from the Neurolaryngology Subcommittee of the American Academy of Otolaryngology-Head and Neck Surgery. Otolaryngol Head Neck Surg. 2007 Jun;136(6):873-81. doi: 10.1016/j.otohns.2007.02.032. PMID 17547973
- [Background] Hamdy S, Aziz Q, Rothwell JC, Crone R, Hughes D, Tallis RC, Thompson DG. Explaining oropharyngeal dysphagia after unilateral hemispheric stroke. Lancet. 1997 Sep 6;350(9079):686-92. doi: 10.1016/S0140-6736(97)02068-0. PMID 9291902
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Smithard DG, O'Neill PA, Parks C, Morris J. Complications and outcome after acute stroke. Does dysphagia matter? Stroke. 1996 Jul;27(7):1200-4. doi: 10.1161/01.str.27.7.1200. PMID 8685928
- [Background] Shaker R, Easterling C, Kern M, Nitschke T, Massey B, Daniels S, Grande B, Kazandjian M, Dikeman K. Rehabilitation of swallowing by exercise in tube-fed patients with pharyngeal dysphagia secondary to abnormal UES opening. Gastroenterology. 2002 May;122(5):1314-21. doi: 10.1053/gast.2002.32999. PMID 11984518
- [Background] Shaker R, Kern M, Bardan E, Taylor A, Stewart ET, Hoffmann RG, Arndorfer RC, Hofmann C, Bonnevier J. Augmentation of deglutitive upper esophageal sphincter opening in the elderly by exercise. Am J Physiol. 1997 Jun;272(6 Pt 1):G1518-22. doi: 10.1152/ajpgi.1997.272.6.G1518. PMID 9227489
- [Background] Logemann JA. Treatment of oral and pharyngeal dysphagia. Phys Med Rehabil Clin N Am. 2008 Nov;19(4):803-16, ix. doi: 10.1016/j.pmr.2008.06.003. PMID 18940642
- [Background] Shaker R, Geenen JE. Management of Dysphagia in stroke patients. Gastroenterol Hepatol (N Y). 2011 May;7(5):308-32. No abstract available. PMID 21857832
- [Background] Easterling C, Grande B, Kern M, Sears K, Shaker R. Attaining and maintaining isometric and isokinetic goals of the Shaker exercise. Dysphagia. 2005 Spring;20(2):133-8. doi: 10.1007/s00455-005-0004-2. PMID 16172822
- [Background] Logemann JA, Rademaker A, Pauloski BR, Kelly A, Stangl-McBreen C, Antinoja J, Grande B, Farquharson J, Kern M, Easterling C, Shaker R. A randomized study comparing the Shaker exercise with traditional therapy: a preliminary study. Dysphagia. 2009 Dec;24(4):403-11. doi: 10.1007/s00455-009-9217-0. Epub 2009 May 27. PMID 19472007
- [Background] Kahrilas PJ, Logemann JA, Krugler C, Flanagan E. Volitional augmentation of upper esophageal sphincter opening during swallowing. Am J Physiol. 1991 Mar;260(3 Pt 1):G450-6. doi: 10.1152/ajpgi.1991.260.3.G450. PMID 2003609